CLINICAL TRIAL: NCT04010708
Title: Iodine Status Monitoring in PortUguese Pregnant woMen: Impact of Supplementation
Acronym: IOMUM
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: NOVA Medical School (Other); Centro Hospitalar De São João, E.P.E. (Other); Hospital de Braga (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: IOMUM
Record Dates: First submitted 2018-08-03; First posted 2019-07-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2019-07

CONDITIONS: Iodine Status in Pregnancy; Iodine Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IOMUM: Pregnant women
  Interventions: Diagnostic Test: Urinary Iodine Concentration Measurement

INTERVENTIONS:
Diagnostic Test: Urinary Iodine Concentration Measurement — UIC

SUMMARY:
Data from 2007 regarding iodine status among Portuguese pregnant women indicate this is an iodine deficient population group, with only 16.8% presenting adequate urinary iodine values. This may have serious implications for normal cognitive development of the offspring and a concerning socioeconomic impact. In 2013, concerns by the Portuguese Directorate-General of Health lead to the implementation of a public health policy (nº 011/2013) recommending iodine supplementation during pregnancy. IoMum emerges from this context to monitor and update iodine status in Portuguese pregnant women and to evaluate the effectiveness of the above policy by assessing clinical compliance to iodine supplementation and the impact of iodine supplementation in this vulnerable group. IoMum will update data on iodine nutrition in Portuguese pregnant women, promoting political actions towards the elimination of iodine deficiency and thus to the reduction of nutritional, social and economic inequalities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the 1st trimester fetal ultrasound scan, from the 10th to the 13th gestational week.

Exclusion Criteria:

* Use of Levothyroxine.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only pregnant women included
Study Population: Portuguese pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
1st trimester urinary iodine concentration | Between gestational weeks 10 and 13 plus 6 days (one timepoint collection - Timepoint 1)
  Median urinary iodine concentration at 1st trimester of gestation
Rate of compliance to iodine supplementation guideline | Between gestational weeks 10 and 13 plus 6 days (one timepoint collection - Timepoint 1)
  Rate of compliance to iodine supplementation guideline at 1st trimester of gestation

SECONDARY OUTCOMES:
Change in median iodine-to-creatinine ratio | Up to 31 weeks
  Change in median iodine-to-creatinine ratio between 1st and 3rd trimesters of gestation
Proportion of pregnant women with insufficient, adequate or excessive iodine intake | Between gestational weeks 10 and 13 plus 6 days (one timepoint collection - Timepoint 1)
  Classification of pregnant women by urinary iodine concentration levels according to WHO criteria (insufficient, adequate or excessive iodine intake) at 1st trimester of gestation.
Maternal median thyroglobulin | Between gestational weeks 35 and 41 (one timepoint collection - Timepoint 2)
  Maternal median thyroglobulin at 3rd trimester of gestation
1st trimester mean sodium excretion | Between gestational weeks 10 and 13 plus 6 days (one timepoint collection - Timepoint 1)
  Mean sodium excretion at 1st trimester of gestation
3rd trimester mean sodium excretion | Between gestational weeks 35 and 41 (one timepoint collection - Timepoint 2)
  Mean sodium excretion at 3rd trimester of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Keating, PhD, Principal Investigator — Center for Health Technology and Services Research; Conceição Calhau, PhD, Principal Investigator — Center for Health Technology and Services Research
Locations (1):
- Faculty of Medicine of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Matta Coelho C, Guimaraes J, Bracchi I, Xavier Moreira N, Pinheiro C, Ferreira P, Pestana D, Barreiros Mota I, Cortez A, Prucha C, Martins C, Pinto E, Almeida A, Delerue-Matos C, Dias CC, Moreira-Rosario A, Ribeiro de Azevedo LF, Cruz Fernandes V, Ramalho C, Calhau C, Brantsaeter AL, Costa Leite J, Keating E. Noncompliance to iodine supplementation recommendation is a risk factor for iodine insufficiency in Portuguese pregnant women: results from the IoMum cohort. J Endocrinol Invest. 2022 Oct;45(10):1865-1874. doi: 10.1007/s40618-022-01813-7. Epub 2022 May 30. PMID 35635644